CLINICAL TRIAL: NCT07197736
Title: Deep Learning for Echo Analysis, Tracking, and Evaluation Prospective Evaluation (DELINEATE-Prospective)
Brief Title: DELINEATE-Prospective
Acronym: DELINEATE
Status: Not yet recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Pierre Elias, Assistant Professor of Medicine in the Department of Biomedical Informatics, Columbia University
Other Study IDs: AAAU9603
Record Dates: First submitted 2025-08-14; First posted 2025-09-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Valve Disease, Aortic; Mitral Regurgitation (MR); Aortic Stenosis; Valvular Heart Disease; Tricuspid Regurgitation (TR); Aortic Regurgitation
Keywords: artificial intelligence; deep learning; valvular heart disease; echocardiography; cardiovascular disease; mitral regurgitation; aortic stenosis
MeSH Terms: conditions — Aortic Valve Disease; Mitral Valve Insufficiency; Aortic Valve Stenosis; Heart Valve Diseases; Tricuspid Valve Insufficiency; Aortic Valve Insufficiency; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: Studies meeting the following criteria will undergo adjudication by an expert panel: Moderate, moderate-severe, or severe mitral, aortic, or tricuspid regurgitation by physician or AI model assessment.
  Discrepancy between physician and AI interpretations, where AI-assessed severity is greater than the physician-assessed severity (i.e. indicates that more valvular regurgitation is present)
- Control Group: A stratified random sample of cases will be selected to match the distribution of AI-flagged cases by physician-assessed valvular regurgitation severity and will undergo the same expert panel adjudication.

SUMMARY:
Heart disease is the leading cause of death in the United States, and echocardiography (or "echo") is the most common way doctors look at the heart. Echo is safe, painless, and can detect major heart problems, including weak heart pumping and valve disease.

Valve disease, especially aortic stenosis (narrowing) and mitral regurgitation (leakage), is common in older adults but often goes undiagnosed. While echo is the main tool for finding valve problems, it takes time, requires expert training, and results can vary between readers.

Recent advances in artificial intelligence (AI), especially deep learning (DL), have shown promise in automatically analyzing heart images. However, past research hasn't fully tackled key echo techniques-like color Doppler and spectral Doppler-that are crucial for measuring how blood moves through heart valves. AI tools also face challenges in being used in everyday medical practice because of workflow issues, lack of real-world testing, and concerns about how the algorithms make decisions.

At Columbia University Irving Medical Center, researchers have built a large database of heart tests over the last six years and developed AI programs to analyze echocardiograms. The current study will test whether providing AI analysis to cardiologists in real time during echo reading can make the process faster and more consistent.

DETAILED DESCRIPTION:
In a prior Columbia University study, a series of deep learning algorithms analyzing echocardiograms is in development. These algorithms include, but are not limited to, algorithms that enable view classification, structure identification, left ventricle (LV) dimension measurements, Left Ventricular Ejection Fraction (LVEF) determination, left atrium (LA) volume assessments, and valvular heart disease diagnosis. Briefly, these algorithms are based on architectures shown to be useful in image and video analysis, including ones specific to echocardiography interpretation. Algorithms based off these architectures can be generalized to interpretation of video-based echocardiogram data such as valvular regurgitation assessment. As part of this study protocol, these models will continue to be developed using patient echocardiogram data. This study aims to create an automated, end-to-end system that can deliver deep learning analyses of echocardiograms to the interpreting cardiologist in real-time. If successful, this program could enable improvements in echocardiography reading efficiency and reliability.

ELIGIBILITY:
Inclusion Criteria:

* Attending cardiologist employed by Columbia University, ColumbiaDoctors, or NewYork Presbyterian Hospital who reads transthoracic echocardiograms in the Columbia echocardiography laboratory
* Provided informed consent to take part in the questionnaires or pivotal study

Exclusion Criteria:

* Physician in training (cardiology fellow or advanced imaging fellow)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Board-certified attending cardiologists at Columbia University, ColumbiaDoctors, or NewYork-Presbyterian Hospital who interpret transthoracic echocardiograms in the Columbia echocardiography laboratory and have provided informed consent to participate
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Clinically Meaningful Reclassification by Panel Review | 18 months
  Proportion of cases where the expert panel reclassifies valvular regurgitation severity by at least one grade (upgrade or downgrade). The proportion will be calculated as the number of cases with reclassification ÷ total number of cases reviewed.

SECONDARY OUTCOMES:
Proportion of Cases with AI-Based Reclassification Leading to a Change in Clinical Management | 18 months
  The proportion will be calculated as the number of cases with any management change ÷ total number of cases reviewed.
Proportion of Cases with AI-Based Reclassification Leading to Referral to a Valve Specialist or Surgeon | 18 months
  Definition: The proportion will be calculated as the number of cases referred to a valve specialist or surgeon ÷ total number of cases reviewed.
Proportion of Cases with AI-Based Reclassification Leading to a Change in Frequency of Follow-Up Echocardiography | 18 months
  The proportion will be calculated as the number of cases with a change in recommended follow-up echocardiography frequency ÷ total number of cases reviewed.
Proportion of Cases with AI-Based Reclassification Leading to Referral for Further Testing (TEE or Cardiac MRI) | 18 months
  The proportion will be calculated as the number of cases referred for further testing with TEE or cardiac MRI ÷ total number of cases reviewed.

OTHER OUTCOMES:
Concordance Between AI and Panel Review | 18 months
  Proportion of cases where AI classification agrees with expert panel review of valvular regurgitation severity.
Concordance Between Cardiologist Clinical Read and Panel Review | 18 months
  Proportion of cases where cardiologist clinical interpretation agrees with expert panel review of valvular regurgitation severity.
Comparison of Concordance Rates (AI vs Cardiologist) Against Panel Review | 18 months
  Difference between the concordance rate of AI vs panel review and the concordance rate of cardiologist clinical read vs panel review.
Inter-Reader Agreement for Categorical Echocardiographic Measures | 18 months
  Agreement between independent cardiologist readers for categorical variables (e.g., severity of valvular regurgitation) will be quantified using Cohen's kappa statistic.
Inter-Reader Agreement for Continuous Echocardiographic Measures | 18 months
  Agreement between independent cardiologist readers for continuous measures (e.g., left ventricular ejection fraction [LVEF] category) will be quantified using the intraclass correlation coefficient (ICC)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre A Elias, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Patient privacy and confidentiality: Even with de-identification, sharing detailed health data could risk re-identification of participants.
  Regulatory restrictions: Institutional Review Boards (IRBs), HIPAA rules, or local laws may limit data sharing, especially for sensitive health information like echocardiograms.
  Consent limitations: If participants did not explicitly consent to broad data sharing at enrollment, the study cannot ethically or legally provide their IPD.